CLINICAL TRIAL: NCT03040856
Title: The Effect of Alpha Linolenic Acid (ALA) Supplementation on Essential Fatty Acids Profile During Pregnancy Compared to Common Supplements and the Epigenetic Effect on the Newborn
Brief Title: The Effect of Alpha Linolenic Acid (ALA) Supplementation During Pregnancy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems executing the study
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Aya Mohr-Sasson, Principal Investigator, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3503-16-SMC
Record Dates: First submitted 2017-02-01; First posted 2017-02-02 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Omega 3 Supplements During Pregnancy
Keywords: Omega 3; Supplements; Alpha Linolenic Acid
MeSH Terms: interventions — alpha-Linolenic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Alpha Linolenic Acid enriched diet (Experimental): Enriched diet with 2 capsules of ALA supplementation a day - 630 mg in each capsule. Total amount of 1260 mg (Daily recommended dose is 1-2 g).
  Interventions: Dietary Supplement: Alpha Linolenic Acid
- Omega 3 enriched diet ( DHA+EPA) (Experimental): Enriched diet with 2 capsules of DHA+EPA supplementation a day (Each capsule consist of 240 mg DHA and 360 mg EPA).
  Interventions: Dietary Supplement: Omega 3 enriched diet ( DHA+EPA)
- Placebo (Placebo Comparator): Control group - Will receive 2 placebo capsule a day - containing olive oil
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Alpha Linolenic Acid — Alpha Linolenic Acid enriched diet
  Arms: Alpha Linolenic Acid enriched diet
Dietary Supplement: Omega 3 enriched diet ( DHA+EPA) — Omega 3 (DHA+EPA) supplementation enriched diet
  Arms: Omega 3 enriched diet ( DHA+EPA)
Other: Placebo — Placebo capsules containing olive oil
  Arms: Placebo

SUMMARY:
Omega-3 fatty acids are "good fats," and are among the most important nutrients lacking in Western diets today. The average person in developing countries consumes less than 100 mg of DHA daily. With increasing awareness of the importance of DHA, many people realize that they need to make a change in their diet by adding DHA-rich foods or supplements.

The aim of this study is to learn the effect of different supplementations from the omega 3 group on the maternal and fetal fatty acid profile during pregnancy and to study their epigenetic influence.

DETAILED DESCRIPTION:
DHA (Docosahexaenoic Acid ) is a long chain omega-3 fatty acid important for brain and eye development and function throughout life. It also supports heart health. DHA is the most abundant omega-3 in the brain and retina and is naturally found in breast milk. EPA (Eicosapentaenoic Acid ) is a long-chain omega-3 fatty acid important for overall health. However, unlike DHA, the body does not store EPA in significant quantities in the brain or retina (DHA is found in every cell throughout the body, EPA is not). These Omega 3 fatty acids are considered essential due to the inability of the human body to create them and the need to consume them from nutritional source. Food that is considered rich in omega 3 fatty acids are fat fish and green vegetables. Omega-3 fatty acids are "good fats," and are among the most important nutrients lacking in Western diets today. The average person in developing countries consumes less than 100 mg of DHA daily. With increasing awareness of the importance of DHA, many people realize that they need to make a change in their diet by adding DHA-rich foods or supplements.

Alpha Linolenic Acid (ALA) is a shorter-chain omega-3 that serves as a source of energy and as a building block for long-chain omega-3 fatty acids (DHA and EPA). This precursor for omega 3 fatty acid is abundant in falx seeds. The mother and the fetus has the metabolic mechanism that enables them to transform ALA into EPA,DHA endogenously.

Women during pregnancy are predisposed to a reduction in unsaturated long chain fatty acid (Polyunsaturated Fatty Acid = PUFA) from the omega 3 group . Lately, a new hypothesis claiming that a reduced level of this essential acids expose the fetus later in his adult life to a spectrum of metabolic and cardiovascular disease. New publication on animal models showed higher rates of obesity, insulin resistance diabetes and cardiovascular damage on mice exposed short chain fatty acids compared to those treated with enriched ALA diet supplementation. Different nutritional and gynecological health organization around the world including the FDA, recommend incorporating omega 3 fatty acids supplementation to daily diet and specifically in pregnant women in order to raise their blood levels for the developing fetus. However, normal fatty acid profile of the omega 3 group in mother and fetus haven't been described yet. Furthermore, the total effect and future benefit to fetus haven't been thoroughly studied and is based mainly on presumptions.

The aim of this study is to learn the effect of different supplementations from the omega 3 group on the maternal and fetal fatty acid profile during pregnancy and to study their epigenetic influence.

Study methods:

Women 12 weeks of gestation visiting high risk unit and fitting inclusion criteria will be offered to participate in the study. Demographic, medical and obstetrical information will be collected from medical files after giving signed informed consent .

Each participant will be randomly assigned to one of three arms of the study based on the order of being recruited (1- to first group, 2- to second group, 3 - to third group, 4- to first group, etc.). Randomization will be done by the principal investigator that is not one of the high risk unit team, and will be blinded to the participants and the treating doctor.

Group 1: Enriched diet with 2 capsules of ALA supplementation a day - 630 mg in each capsule. Total amount of 1260 mg (Daily recommended dose is 1-2 g).

Group 2: Enriched diet with 2 capsules of DHA+EPA supplementation a day (Each capsule consist of 240 mg DHA and 360 mg EPA) Group 3: Control group - Will receive 2 placebo capsule a day (All products will be supplied by the same company that is approved by the FDA and the Israeli health ministry) Follow up will take place on every visit to the high risk unit that is 3 and 2 weeks apart at the second and third trimester, respectively. On each visit one blood tube that include 5cc of blood will be taken for fatty acid profile analysis and on labor 2 blood tubes will be taken from the mother and from the umbilical cord after separation of the placenta : 1- for fatty acid analysis , 2- for PCR evaluation of mRNAs of genes that were found correlated in animal models to be influenced by maternal diet during pregnancy and are connected to metabolic syndrome pathologies in adulthood ( including - FASn, Elov6, PPAR (α, β/δ, γ), SCD1, Fads2, SREBP-1 Ppargc1alpha, Lpin1, Plin5 , MAPK/PGC-1α. (

ELIGIBILITY:
Inclusion Criteria:

* Age 18-42
* Singleton
* Gestational age 12-16 during first visit at the high risk unit

Exclusion Criteria:

* Liver Disease
* Dyslipidemia
* Twins
* Warfarin, LMWH, Heparin use ( Due to suspected drug interaction that has been reported however has not been proven yet)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 0 (Actual)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Levels of Omega 3 fatty acids ( DHA, EPA, ALA) | Change in maternal levels of Omega 3 fatty acids ( DHA, EPA, ALA) from recruitment (12 week of gestation ) until delivery .
  Change in Omega 3 fatty acids ( DHA, EPA, ALA) blood levels during different gestational weeks of pregnancy until delivery, including umbilical cord blood levels after the separation of the placenta ( third stage of delivery).

SECONDARY OUTCOMES:
Expression of messenger RNAs ( mRNAs) between the study groups | At delivery - Immediately after separation of the placenta ( Blood sample from the mother and from the umbilical cord)
  Change between study groups in expression of mRNAs in the mother at delivery and in the fetus ( analyzing umbilical cord blood after separation of the placenta) ( including - FASn, Elov6, PPAR (α, β/δ, γ), SCD1, Fads2, SREBP-1 Ppargc1alpha, Lpin1, Plin5 , MAPK/PGC-1α)

CONTACTS AND LOCATIONS:
Overall Officials: Israel Hendler, M.D, Study Director — Department of Obstetrics and Gynecology ,Sheba Medical Center, Ramat Gan, Israel; Alicia Leikin-Frenkel, M.D, Ph.d, Study Director — Bert Strassburger Lipid Center, Sheba Medical Center, Ramat Gan, Israel
Locations (1):
- Dr. A Mohr-Sasson, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu JC, Raine A, Ang RP, Fung DS. An analysis of blinding success in a randomised controlled trial of fish oil omega-3 fatty acids. Ann Acad Med Singap. 2015 Mar;44(3):85-91. PMID 25882235
- [Result] Grey A, Bolland M. Clinical trial evidence and use of fish oil supplements. JAMA Intern Med. 2014 Mar;174(3):460-2. doi: 10.1001/jamainternmed.2013.12765. No abstract available. PMID 24352849
- [Result] Tsyb AF, Parshkov EM, Sokolov VA. [Major trends of research at the Research Institute of Medical Radiology of the USSR Academy of Medical Sciences under the 12th 5-Year Plan]. Med Radiol (Mosk). 1987 Sep;32(9):6-10. No abstract available. Russian. PMID 3657456
- [Result] Hure A, Young A, Smith R, Collins C. Diet and pregnancy status in Australian women. Public Health Nutr. 2009 Jun;12(6):853-61. doi: 10.1017/S1368980008003212. Epub 2008 Jul 23. PMID 18647425
- [Result] Diet, nutrition and the prevention of chronic diseases. World Health Organ Tech Rep Ser. 2003;916:i-viii, 1-149, backcover. PMID 12768890
- [Result] Kris-Etherton PM, Innis S, Ammerican Dietetic Assocition, Dietitians of Canada. Position of the American Dietetic Association and Dietitians of Canada: dietary fatty acids. J Am Diet Assoc. 2007 Sep;107(9):1599-611. PMID 17936958
- [Result] Harris WS, Mozaffarian D, Lefevre M, Toner CD, Colombo J, Cunnane SC, Holden JM, Klurfeld DM, Morris MC, Whelan J. Towards establishing dietary reference intakes for eicosapentaenoic and docosahexaenoic acids. J Nutr. 2009 Apr;139(4):804S-19S. doi: 10.3945/jn.108.101329. Epub 2009 Feb 25. PMID 19244379
- [Result] Innis SM. Essential fatty acid transfer and fetal development. Placenta. 2005 Apr;26 Suppl A:S70-5. doi: 10.1016/j.placenta.2005.01.005. PMID 15837071
- [Result] Weaver KL, Ivester P, Seeds M, Case LD, Arm JP, Chilton FH. Effect of dietary fatty acids on inflammatory gene expression in healthy humans. J Biol Chem. 2009 Jun 5;284(23):15400-7. doi: 10.1074/jbc.M109.004861. Epub 2009 Apr 9. PMID 19359242
- [Result] Casanova MA, Medeiros F, Trindade M, Cohen C, Oigman W, Neves MF. Omega-3 fatty acids supplementation improves endothelial function and arterial stiffness in hypertensive patients with hypertriglyceridemia and high cardiovascular risk. J Am Soc Hypertens. 2017 Jan;11(1):10-19. doi: 10.1016/j.jash.2016.10.004. Epub 2016 Oct 26. PMID 27876342
- [Result] Shomonov-Wagner L, Raz A, Leikin-Frenkel A. Alpha linolenic acid in maternal diet halts the lipid disarray due to saturated fatty acids in the liver of mice offspring at weaning. Lipids Health Dis. 2015 Feb 26;14:14. doi: 10.1186/s12944-015-0012-7. PMID 25889505
- [Result] Hollander KS, Tempel Brami C, Konikoff FM, Fainaru M, Leikin-Frenkel A. Dietary enrichment with alpha-linolenic acid during pregnancy attenuates insulin resistance in adult offspring in mice. Arch Physiol Biochem. 2014 Jul;120(3):99-111. doi: 10.3109/13813455.2014.940352. Epub 2014 Jul 17. PMID 25030769
- [Result] Leikin-Frenkel AI. Is there A Role for Alpha-Linolenic Acid in the Fetal Programming of Health? J Clin Med. 2016 Mar 23;5(4):40. doi: 10.3390/jcm5040040. PMID 27023621
- [Result] Leikin-Frenkel A, Shomonov-Wagner L, Juknat A, Pasmanik-Chor M. Maternal Diet Enriched with alpha-Linolenic or Saturated Fatty Acids Differentially Regulates Gene Expression in the Liver of Mouse Offspring. J Nutrigenet Nutrigenomics. 2015;8(4-6):185-94. doi: 10.1159/000442945. Epub 2016 Jan 21. PMID 26788914
- [Result] Leikin-Frenkel A, Goldiner I, Leikin-Gobbi D, Rosenberg R, Bonen H, Litvak A, Bernheim J, Konikoff FM, Gilat T. Treatment of preestablished diet-induced fatty liver by oral fatty acid-bile acid conjugates in rodents. Eur J Gastroenterol Hepatol. 2008 Dec;20(12):1205-13. doi: 10.1097/MEG.0b013e3282fc9743. PMID 18989145